CLINICAL TRIAL: NCT01550016
Title: Clinical Evaluation of Dengue and Identification of Risk Factors for Severe Disease (WP1)
Brief Title: International Research Consortium on Dengue Risk Assessment, Management, and Surveillance
Acronym: IDAMS
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: European Union (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Thomas Jaenisch, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: 281803 (EU FP7-HEALTH-2011)
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Dengue Fever
Keywords: dengue warning signs; latin america; south east asia; other febrile illnesses; dengue classification
MeSH Terms: conditions — Dengue | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Febrile Patients: Observation of patients with possible dengue fever in the early phase of disease
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Clinical follow-up and laboratory investigations.

SUMMARY:
Improvements in diagnosis of dengue fever and prediction of which patients will get more severe disease are urgently needed to improve the treatment of patients with dengue. This is very important in places with many people who suffer from dengue but have limited health care resources. This study will enroll patients with fever which may be caused by dengue in 6 countries with high incidence of dengue over two continents (Brazil, Cambodia, El Salvador, Indonesia, Malaysia and Vietnam). All patients will be followed by a doctor with blood tests and exams until they recover. Symptoms and laboratory tests will be followed so that the cause of fever can be determined. For patients who have dengue, the investigators will look for symptoms and tests which indicate more serious disease. This study will help to determine how to identify patients with dengue fever based on symptoms and simple laboratory tests and those who will get more serious disease. It will also help to define a more standardized management of patients with dengue fever.

DETAILED DESCRIPTION:
Improvements in clinical diagnosis of dengue and risk prediction for severe disease are urgently needed to improve overall clinical care, especially in settings with a high case burden where appropriate allocation of limited resources is crucial to outcome. In this work package 10,000 outpatients with undifferentiated fever, consistent with possible dengue, will be recruited within 3 days of fever onset in 6 endemic countries (Brazil, Cambodia, El Salvador, Indonesia, Malaysia and Vietnam), and will be followed daily until full recovery. Clinical features and simple laboratory parameters differentiating dengue from other febrile illness will be identified, and, among those with confirmed dengue, risk factors for progression to more severe disease will be evaluated. As well as contributing to the development of diagnostic and prognostic algorithms the clinical cohort has considerable potential towards standardisation of procedures for dengue management and reporting.

ELIGIBILITY:
Inclusion Criteria:

* >= 5 years of age
* fever for less than 72 hours

Exclusion Criteria:

* presence of localizing signs suggestive of another diagnosis
* not likely to come back for daily follow-up
* complications or signs of severe disease

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Febrile patients presenting to outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 7411 (Actual)
Dates: Start 2011-10; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Hospitalization or administration of IV fluid | 14 days
  Proportion of dengue patients hospitalized or treated with IV fluids within 14 days of enrollment.

SECONDARY OUTCOMES:
Development of severe disease | 14 days
  Development of severe disease according to the 2009 WHO Dengue classification within 14 days of enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jänisch, Principal Investigator — Heidelberg University Medical Center
Locations (9):
- International Centre for Diarrhoeal Diseases, Dhaka, Dhaka Division, Bangladesh
- Brazil (2):
  - Fundacao Oswaldo Cruz (FIOCRUZ), Rio de Janeiro, Rio de Janeiro
  - Fundacao Universidade Estadual do Ceara, Fortaleza
- Angkor Hospital for Children, Siem Reap, Cambodia
- Hospital National de Ninos Benjamin Bloom, San Salvador, El Salvador
- Gadjah Madah University, Yogyakarta, Indonesia
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia
- Universidad de Carabobo, Valencia, Valencia, Venezuela
- Oxford University Clinical Research Unit, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaenisch T, Tam DT, Kieu NT, Van Ngoc T, Nam NT, Van Kinh N, Yacoub S, Chanpheaktra N, Kumar V, See LL, Sathar J, Sandoval EP, Alfaro GM, Laksono IS, Mahendradhata Y, Sarker M, Ahmed F, Caprara A, Benevides BS, Marques ET, Magalhaes T, Brasil P, Netto M, Tami A, Bethencourt SE, Guzman M, Simmons C, Quyen NT, Merson L, Dung NT, Beck D, Wirths M, Wolbers M, Lam PK, Rosenberger K, Wills B. Clinical evaluation of dengue and identification of risk factors for severe disease: protocol for a multicentre study in 8 countries. BMC Infect Dis. 2016 Mar 11;16:120. doi: 10.1186/s12879-016-1440-3. PMID 26968374
- See also: IDAMS consortium — http://www.idams.eu
- See also: Section Clinical Tropical Medicine, Heidelberg University Medical Center, Germany — http://www.klinikum.uni-heidelberg.de/Sektion-Klinische-Tropenmedizin.5489.0.html
- See also: Oxford University Clinical Research Unit, Viet Nam — http://www.oucru.org